CLINICAL TRIAL: NCT00050895
Title: A Phase III, Randomized, Open-Label Comparison of Lopinavir/Ritonavir Plus Efavirenz Versus Lopinavir/Ritonavir Plus 2 NRTIs Versus Efavirenz Plus 2 NRTIs as Initial Therapy for HIV-1 Infection
Brief Title: Comparing the Safety, Effectiveness, and Tolerability of Three Anti-HIV Drug Regimens for Treatment-Naive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5142; 10085 (Registry Identifier: DAIDS ES); ACTG A5142; A5152s; A5160s
Record Dates: First submitted 2002-12-30; First posted 2003-01-01 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Reverse Transcriptase Inhibitors; HIV Protease Inhibitors; Drug Therapy, Combination; Delayed Action Preparations; Treatment Naive; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; efavirenz; Stavudine; Zidovudine; Lamivudine; Tenofovir

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Efavirenz
Drug: Stavudine
Drug: Zidovudine
Drug: Lamivudine
Drug: Tenofovir disoproxil fumarate

SUMMARY:
With new strategies and drugs available, many different regimens exist for the treatment of HIV. The purpose of this study is to compare three different anti-HIV drug regimens as first-time treatments for HIV infection.

DETAILED DESCRIPTION:
Numerous treatment options are available to HIV infected patients who are antiretroviral (ARV) therapy naive, but an optimal regimen has not yet been established. This study will compare a nonnucleoside reverse transcriptase inhibitor (NNRTI)-based regimen, a ritonavir (RTV)-enhanced protease inhibitor (PI)-based regimen, and a nucleoside reverse transcriptase inhibitor (NRTI)-sparing regimen for the initial treatment of HIV infection.

Patients will be randomly assigned to one of three study arms. In Arm A, patients will receive lopinavir/ritonavir (LPV/r) twice daily and efavirenz (EFV) once daily before bed. Arm B patients will receive LPV/r twice daily, lamivudine (3TC) once daily, plus either stavudine extended release (d4T XR) once daily, zidovudine (ZDV) twice daily, or tenofovir disoproxil fumarate (TDF) once daily. Patients in Arm C will receive EFV once daily before bed and 3TC plus either d4T XR once daily before bed, ZDV twice daily, or TDF once daily before bed.

Study visits will occur every 4 weeks until Week 24, then every 8 weeks thereafter for a maximum of 96 weeks. Blood will be drawn at every visit and a urine sample will be collected every 8 weeks. Body measurements will be taken at Weeks 24, 48, 72, and 96. Whole body dual-energy x-ray absorptiometry (DEXA) scans will be done at Weeks 48 and 96. Patients must fast before study visits at Weeks 12, 24, 48, 72, and 96. Women in the study will have gynecological assessments every 24 weeks.

ELIGIBILITY:
Inclusion Criteria for Step 1:

* HIV infected
* HIV viral load of 2000 copies/ml or greater within 60 days prior to study entry
* Willing to use acceptable means of contraception
* d4T XR, TDF, or ZDV chosen as part of an initial regimen prior to randomization to a study arm
* Coenrolled in ACTG A5152s

Exclusion Criteria for Step 1:

* On ARV therapy for 7 days or more any time prior to study entry
* NNRTIs or 3TC at any time prior to study entry
* Current peripheral neuropathy of Grade 2 or higher
* Pregnancy or breastfeeding
* Immunomodulators, vaccines, or investigational therapies within 30 days of study entry. Patients taking a stable or tapering dose of prednisone at less than 10 mg are not excluded.
* Human growth hormone within 30 days prior to study entry
* Initiation of testosterone or anabolic steroids within 30 days prior to study entry
* Certain other medications within 30 days of study entry
* Hypersensitivity to components of the study drug formulations
* Drug or alcohol use or dependence that would interfere with adherence to study requirements
* Acute therapy for serious medical illnesses requiring systemic treatment and/or hospitalization within 14 days prior to study entry
* Recent infection with drug-resistant HIV

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 775
Dates: Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time from study entry to virologic failure
time from study entry to regimen completion

SECONDARY OUTCOMES:
20 % or more loss in peripheral fat
increase in lactic acid levels at least 2-4old above the upper limit of normal (ULN)
20 % or more increase in truncal fat accumulation
fasting cholesterol level equal to or greater than 240 mg/dl
Grade 3 or greater elevation in fasting triglyceride levels
change from baseline in insulin resistance | at Weeks 24, 48 and 96
change from baseline of whole-body bone density and whole-body bone mineral content | at Weeks 48 and 96
time to confirmed virologic failure while on Steps I (initial randomized regimen) or II (within class substitutes for initial regimen toxicity) OR treatment-limiting toxicity on Steps I or II
number of antiretroviral classes with resistance mutations at virologic failure
number of missed medication doses | 4 days prior
change from baseline in self-reported symptoms OR occurrence of reporting an increase in symptoms | at Weeks 4, 48, 72 and 96
change from baseline in body image OR occurrence of reporting body image distress | at Weeks 24, 48, 72 and 96
time until treatment-limiting toxicity OR occurrence of Grades 3 or 4 toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Riddler, MD, Study Chair — University of Pittsburgh; Richard Haubrich, MD, Study Chair — University of California, San Diego, Division of Infectious Diseases
Locations (60):
- United States (59):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Indiana Univ. School of Medicine, Wishard Memorial, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - SSTAR, Family Healthcare Ctr., Fall River, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell CRS, New York, New York
  - Columbia Univ., HIV Prevention and Treatment Medical Ctr., New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - AIDS Care CRS, Rochester, New York
  - McCree McCuller Wellness Ctr. at the Connection, Infectious Disease Unit, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Wake County Health and Human Services CRS, Raleigh, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Cleveland Clinic Foundation, Div. of Medicine, Infectious Diseases, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - Rhode Island Hosp., Providence, Rhode Island
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington
- Durban Adult HIV CRS, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Background] Saint-Marc T, Partisani M, Poizot-Martin I, Rouviere O, Bruno F, Avellaneda R, Lang JM, Gastaut JA, Touraine JL. Fat distribution evaluated by computed tomography and metabolic abnormalities in patients undergoing antiretroviral therapy: preliminary results of the LIPOCO study. AIDS. 2000 Jan 7;14(1):37-49. doi: 10.1097/00002030-200001070-00005. PMID 10714566
- [Background] DiRienzo AG, DeGruttola V. Design and analysis of clinical trials with a bivariate failure time endpoint, with application to AIDS Clinical Trials Group Study A5142. Control Clin Trials. 2003 Apr;24(2):122-34. doi: 10.1016/s0197-2456(02)00321-5. PMID 12689734
- [Result] Von Burg R, Stout T. Paraldehyde. J Appl Toxicol. 1991 Oct;11(5):379-81. doi: 10.1002/jat.2550110515. No abstract available. PMID 1783744
- [Result] Haubrich RH, Riddler SA, DiRienzo AG, Komarow L, Powderly WG, Klingman K, Garren KW, Butcher DL, Rooney JF, Haas DW, Mellors JW, Havlir DV; AIDS Clinical Trials Group (ACTG) A5142 Study Team. Metabolic outcomes in a randomized trial of nucleoside, nonnucleoside and protease inhibitor-sparing regimens for initial HIV treatment. AIDS. 2009 Jun 1;23(9):1109-18. doi: 10.1097/QAD.0b013e32832b4377. PMID 19417580
- [Result] Gazzard B, Balkin A, Hill A. Analysis of neuropsychiatric adverse events during clinical trials of efavirenz in antiretroviral-naive patients: a systematic review. AIDS Rev. 2010 Apr-Jun;12(2):67-75. PMID 20571601
- [Result] Simpson KN, Dietz B, Baran RW, Garren KW, Riddler SA, Bhor M, Haubrich RH. Economic modeling of the combined effects of HIV-disease, cholesterol and lipoatrophy based on ACTG 5142 trial data. Cost Eff Resour Alloc. 2011 May 8;9:5. doi: 10.1186/1478-7547-9-5. PMID 21548986
- [Derived] Cardone KM, Dudek S, Keat K, Bradford Y, Cindi Z, Daar ES, Gulick R, Riddler SA, Lennox JL, Sinxadi P, Haas DW, Ritchie MD. Lymphocyte Count Derived Polygenic Score and Interindividual Variability in CD4 T-cell Recovery in Response to Antiretroviral Therapy. Pac Symp Biocomput. 2024;29:594-610. PMID 38160309
- [Derived] Li B, Veturi Y, Verma A, Bradford Y, Daar ES, Gulick RM, Riddler SA, Robbins GK, Lennox JL, Haas DW, Ritchie MD. Tissue specificity-aware TWAS (TSA-TWAS) framework identifies novel associations with metabolic, immunologic, and virologic traits in HIV-positive adults. PLoS Genet. 2021 Apr 26;17(4):e1009464. doi: 10.1371/journal.pgen.1009464. eCollection 2021 Apr. PMID 33901188
- [Derived] Leonard MA, Cindi Z, Bradford Y, Bourgi K, Koethe J, Turner M, Norwood J, Woodward B, Erdem H, Basham R, Baker P, Rebeiro PF, Sterling TR, Hulgan T, Daar ES, Gulick R, Riddler SA, Sinxadi P, Ritchie MD, Haas DW. Efavirenz Pharmacogenetics and Weight Gain Following Switch to Integrase Inhibitor-Containing Regimens. Clin Infect Dis. 2021 Oct 5;73(7):e2153-e2163. doi: 10.1093/cid/ciaa1219. PMID 32829410
- [Derived] Mollan KR, Smurzynski M, Eron JJ, Daar ES, Campbell TB, Sax PE, Gulick RM, Na L, O'Keefe L, Robertson KR, Tierney C. Association between efavirenz as initial therapy for HIV-1 infection and increased risk for suicidal ideation or attempted or completed suicide: an analysis of trial data. Ann Intern Med. 2014 Jul 1;161(1):1-10. doi: 10.7326/M14-0293. PMID 24979445
- [Derived] Bronke C, Almeida CM, McKinnon E, Roberts SG, Keane NM, Chopra A, Carlson JM, Heckerman D, Mallal S, John M. HIV escape mutations occur preferentially at HLA-binding sites of CD8 T-cell epitopes. AIDS. 2013 Mar 27;27(6):899-905. doi: 10.1097/QAD.0b013e32835e1616. PMID 23276808
- [Derived] Hulgan T, Haubrich R, Riddler SA, Tebas P, Ritchie MD, McComsey GA, Haas DW, Canter JA. European mitochondrial DNA haplogroups and metabolic changes during antiretroviral therapy in AIDS Clinical Trials Group Study A5142. AIDS. 2011 Jan 2;25(1):37-47. doi: 10.1097/QAD.0b013e32833f9d02. PMID 20871389
- [Derived] Riddler SA, Haubrich R, DiRienzo AG, Peeples L, Powderly WG, Klingman KL, Garren KW, George T, Rooney JF, Brizz B, Lalloo UG, Murphy RL, Swindells S, Havlir D, Mellors JW; AIDS Clinical Trials Group Study A5142 Team. Class-sparing regimens for initial treatment of HIV-1 infection. N Engl J Med. 2008 May 15;358(20):2095-106. doi: 10.1056/NEJMoa074609. PMID 18480202